CLINICAL TRIAL: NCT02882906
Title: Myofascial Trigger Points Are Associated in the Upper Limb in Stroke Patients: a Cross Sectional Study
Brief Title: Myofascial Trigger Points in the Upper Limb in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Jorge Hugo Villafañe, PhD, Researcher, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: MTrPs
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Stroke
Keywords: Stroke; Pain; Shoulder
MeSH Terms: conditions — Stroke; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
One source of shoulder pain can be myofascial trigger points (MTrPs). MTrPs are localized, hyperirritable points in the skeletal muscles that are associated with palpable nodules in muscle fibres. MTrPs can be classified into active and latent. Latent MTrPs demonstrate the same clinical characteristics as active MTrPs but they do not provoke spontaneous pain. Numerous studies have shown that MTrPs are prevalent in patients with chronic non-traumatic neck and shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral shoulder pain and a physician-diagnosed stroke.

Exclusion Criteria:

* Rheumatic inflammatory,
* Systemic diseases,
* Acute traumatic conditions,
* Postoperative conditions, neck and elbow disorders, and
* Serious aphasias in which there was a communication problem.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with a complaint of shoulder pain following a stroke were recruited to be subjects in the study following referral to physical therapy to the outpatient department at orthopedic rehabilitation facility by a family practice physician.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change of Pain intensity | Baseline
  Visual Analogue Scale
Pressure Pain Thresholds (PPT) | Baseline
  PPT will be assessed the shoulder Stroke (infraspinatus, supraspinatus, teres minor and upper trapezius).

SECONDARY OUTCOMES:
Barthel index | Baseline
  Barthel index
DASH | Baseline
  The Disabilities of the Arm, Shoulder and Hand Score

CONTACTS AND LOCATIONS:
Overall Officials: JORGE H VILLAFAÑE, PhD, Principal Investigator — IRCCS Don Gnocchi Foundation
Locations (1):
- Jorge Hugo Villafañe, Piossasco, Turin, Italy

IPD SHARING:
Plan to Share IPD: No